CLINICAL TRIAL: NCT04933825
Title: An Exploratory,Open-label,and Single Center Study to Evaluate the Safety and Efficacy of ET-02 in Patients With Relapsed or Refractory B-cell Malignancies(NHL/ALL).
Brief Title: A Study of ET-02 in Patients With Relapsed or Refractory B-cell Malignancy(NHL/ALL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: EdiGene (GuangZhou) Inc. (Industry)
Collaborators: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDI-002
Record Dates: First submitted 2021-06-09; First posted 2021-06-22 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Relapsed or Refractory B-cell Malignancy(NHL/ALL)
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Four escalating dose-levels of ET-02 will be evaluated using a "3+3" design. (Experimental)
  Interventions: Biological: ET-02

INTERVENTIONS:
Biological: ET-02 — A conditioning therapy with cyclophosphamide and fludarabine will be conducted before ET-02 injection.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CD19-UCART in patients with r/r B-cell hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteer to participate in the study and sign the ICF;
2. Male or female aged≥18 years old；
3. Patient with relapsed or refractory CD19 positive B-ALL orNHL，as evidenced by 2 or more lines of prior therapy ;
4. Estimated life expectancy≥12 weeks ;
5. ECOG performance status ≤1;
6. Adequate organ function.

Exclusion Criteria:

1. Patients with graft-versus-host disease (GVHD) or requiring immunosuppressive therapy；
2. History of central nervous system (CNS) involvement by malignancy；
3. Women who are pregnant or breastfeeding；
4. Any situations that may increase the risk of patients or interfere with the results of study，which judged by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 2 years after lymphodepleting chemotherapy
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- •The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China